CLINICAL TRIAL: NCT06815939
Title: Validation of a Lab-free Low-cost Screening Test for Prevention of Cervical Cancer: Automated Visual Evaluation
Brief Title: Validation of a Lab-free Low-cost Screening Test for Prevention of Cervical Cancer
Acronym: OPTICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DL Analytics (Industry)
Collaborators: Basic Health International (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 4R44CA247137 (NIH); 4R44CA247137 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-02-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus (HPV); Cervical Intraepithelial Neoplasia; Uterine Cervical Neoplasms; Cervical Cancers
Keywords: Human Papillomavirus; Cervical Cancer; Screening; Neoplasms; Precancerous Conditions; Uterine Diseases; Uterine Cervical Diseases; Genital Diseases, Female; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Genital Diseases; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Neoplasms; Precancerous Conditions; Uterine Diseases; Uterine Cervical Diseases; Genital Diseases, Female; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Genital Diseases; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site | interventions — Human Papillomavirus DNA Tests; Watchful Waiting; Acetic Acid; Pregnancy Tests; Colposcopy; Biopsy; Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Women eligible for HPV screening based on El Salvador's national guidelines will receive careHPV, VIA, and AVE (active comparator).
  Screen-positive women by HPV, VIA or AVE referred to colposcopy clinic and 5% of screen-negative women (negative on HPV, VIA, and AVE).
  Cervical cancer triage and diagnostic tests among screen- positive women and screen negative women.
  Biopsy-confirmed positive will receive necessary treatment by local standard of care.
  Interventions: Diagnostic Test: HPV Test; Device: EVA System; Procedure: Visual Inspection with Acetic Acid (VIA); Diagnostic Test: Automated Visual Evaluation (AVE); Other: Image Capture with Mobile Phone; Diagnostic Test: Pregnancy test; Diagnostic Test: ScreenFire HPV test; Procedure: Colposcopy with biopsy; Procedure: Thermal Ablation; Procedure: Loop electrosurgical excision procedure (LEEP)

INTERVENTIONS:
Diagnostic Test: HPV Test — The careHPV (QIAGEN, Gaithersburg, MD) test was developed in a public-private partnership specifically for use in low-resource settings. It is a simplified, robust, and affordable HPV test that does not distinguish specific HPV types; rather, it gives a positive result if any of 14 hrHPV types is present in the specimen. Electricity is necessary to run the test, but it does not need running water or air conditioning. In order to be most cost effective, the samples must be run with a full plate of 96 samples. Results take 3-4 hours to complete.
Device: EVA System — Digital colposcope
Procedure: Visual Inspection with Acetic Acid (VIA) — unaided visual inspection with acetic acid
Diagnostic Test: Automated Visual Evaluation (AVE) — Digital diagnostic classification, quality classifier using captured images from EVA System
  Other Names: CINFinder
Other: Image Capture with Mobile Phone — Compare performance of AVE installed on a mobile phone vs. on the EVA System
Diagnostic Test: Pregnancy test — Urine based pregnancy test
Diagnostic Test: ScreenFire HPV test — ScreenFire HPV test (Atila BioSystems, Inc, Mountain View, CA) uses isothermal amplification to detect 13 high risk (hr)HPV types directly from clinical samples in approximately one hour. The test can be run on any real-time PCR machine and gives separate results for hrHPV types 16 and 18, as well as a pooled positive result for 13 other hrHPV types. The human cellular gene beta-globin is used as an internal control to measure sample adequacy. ScreenFire can be self-collected and does not require batching. AmpFire® obtained CE-mark in 2017.
Procedure: Colposcopy with biopsy — A colposcopic exam with biopsy entails visual magnification of the cervix and the removal of a small piece of cervical tissue. After the application of acetic acid 5% onto the cervix, a device called a colposcope allows the clinician to visually identify changes consistent with HPV. Areas of the cervix where lesions appear (or if not, randomly selected sections) are then biopsied (small piece of sample removed) and an endocervical curettage is performed (removing a small section from the inside of the cervix). Tissue specimens are then sent to the lab for pathology diagnosis.
Procedure: Thermal Ablation — Thermal ablation is utilized to treat high-grade cervical precancer. First, a speculum is introduced into the vagina to identify the cervix. Acetic acid 5% is applied to the cervix for one minute and the cervix is observed to look for changes consistent with precancer. If the cervix is able to be fully evaluated and there are no signs of invasive cancer, the tip of the device is heated to 100ºC and applied directly to the cervix for 1-2 minutes, which ablates or destroys the abnormal cells.
Procedure: Loop electrosurgical excision procedure (LEEP) — LEEP is utilized to remove abnormal tissue from the cervix. This may include tissue with precancerous cells (called cervical dysplasia) or cancerous cells. The loop is heated using electricity to remove the tissue. LEEP may also be called a loop excision or large loop excision of the transformation zone (LLETZ).

SUMMARY:
The purpose of this study is to validate Automated Visual Evaluation (AVE), specifically the CINFinder version developed by DL Analytics, a point-of-care screening and triage diagnostic tool for cervical cancer based on the assessment of digital images through artificial intelligence. Several teams around the world have developed versions of AVE as a triage technology but none as a screening tool.

DETAILED DESCRIPTION:
BACKGROUND:

Cervical cancer, caused by persistent infection of carcinogenic types of the human papillomavirus (HPV), is the second leading cause of female cancer in El Salvador. Effective screening and treatment of precancerous lesions have lowered cervical cancer rates in high-income countries, but the disease remains a leading cause of death in low-and middle-income countries (LMICs). Currently, up to 80% of the disease burden and 90% of global deaths occur in LMICs primarily due to lack of resources and poor infrastructure. A new test, Automated Visual Evaluation (AVE), is a point-of-care screening and triage diagnostic tool based on the assessment of digital images through artificial intelligence.

The purpose of this study is to validate Automated Visual Evaluation (AVE), specifically the CINFinder version developed by DL Analytics, a point-of-care screening and triage diagnostic tool based on the assessment of digital images through artificial intelligence. AVE has been in development since 2021. The current study will consist of a clinical trial to compare the sensitivity of AVE (CINFinder version) with traditional screening and triage tests.

STUDY DESIGN:

This is a prospective paired interventional study of 10,000 women in San Salvador, El Salvador, to test the difference in sensitivities between AVE (CINFinder) and with other screening and triage tests, including HPV tests and unaided visual inspection with acetic acid (VIA) to detect CIN2+ as a primary screening method. As a secondary aim, investigators will also validate the use of AVE as a triage test in patients with positive HPV results. Histopathology diagnosis will be used as the reference to determine true disease status.

STUDY PROCEDURES:

The design includes a screening visit, a colposcopy visit, and a result delivery and treatment visit. During the screening visit, participants will undergo routine HPV sample collection, VIA, AVE with the EVA System (digital colposcope), and an additional cervical image capture with an Android smartphone. Women with a positive screening result on any of the three main screening tests (HPV test, VIA, or AVE with the EVA System) will be referred to a second study visit to undergo HPV testing with a genotyping test, AVE with the EVA System for the second time, and colposcopy with biopsy. In addition, 5% of screen-negative women will undergo the same procedures. Results from VIA and AVE with the EVA System during the first and the second visit will be compared to determine AVE performance as a screening and triage test, respectively. Histopathology findings will serve as the reference to establish the true diagnosis of each case. Women will receive their histopathology results during the third visit and, if eligible, will be offered ablation treatment the same day. Women ineligible for ablation will be referred to LEEP or other care as appropriate.

DATA COLLECTION & MANAGEMENT:

This specific version of AVE (CINFinder) is designed to run on both EVA System and an Android phone, alongside additional tools for improving image quality and post-screening management.The AVE software (including CINFinder, CerVisibility, and CervManager modules), will be installed as user-friendly features that can be easily accessed by authorized

Data collection: All data will be recorded in real time on paper forms OR on an electronic tablet filled out by a nurse research assistant. All forms (digital or paper) will include the date and study ID to link information to specific patients and visits. Collected data will include eligibility criteria, a background questionnaire including relevant sociodemographic and medical history traits, clinical procedures, and laboratory results. In addition, providers conducting speculum exams during the first (screening) and second (colposcopy and biopsy) visits will use the CervManager application to create a profile for each patient to input clinical information. Thus, study data will be collected on both paper forms and CervManager for added back-up security. Providers will also capture cervical images using the CervManager application on both the EVA System and an Android mobile phone. Images belonging to the same patient will be synchronized under the same study ID. Other clinical data (e.g., HPV test results, histopathology) will also be inputted into the CervManager patient profile.

Data Management: For storage and management, data from paper forms will be transferred to REDCap, an electronic data management system widely used for clinical research. CervManager and REDCap can be downloaded and merged periodically to easily identify and correct any entry errors, duplications, or missing data on either database. All AVE algorithms implemented as part of this project and used for subsequent analyses will run on DL Analytics servers.

Non-participant documentation: Investigators will document the number of eligible women who decline to participate in the study (including main reasons why). If individuals agree, Investigators will collect general, de-identified information (i.e., age range, education, and previous screening). This will be done to identify any potential source of sampling bias.

STATISTICAL POWER CALCULATIONS AND SAMPLE SIZES

Aim 1: Validate AVE as a primary screening test compared to visual inspection with acetic acid (VIA) for the detection of high-grade cervical pre- cancer (CIN2+).

A study with 10,000 women will be able to detect a minimum difference of 10% between VIA and AVE with 80% power and a Type I error rate of 5%, assuming a minimum sensitivity of VIA of 65% and a correlation coefficient of the tests in the diseased population (Rho) of at least 50%. Based on the study design, all participants who test positive on any test will be referred to colposcopy with biopsy (i.e., proportion of verification = 1), as opposed to only 5% of those who are double negative being referred (i.e., proportion of verification = 0.05). Finally, based on the Investigators previous experience working in El Salvador, Investigators estimate the prevalence (lambda) of CIN2+ in the general screening population at 2%.

Objective 2. To compare AVE as a triage test compared to VIA for detecting CIN2+ among HPV-positive women.

Since all women who test positive with careHPV, VIA or AVE will undergo colposcopy with biopsy, the positive predictive value (PPV) for CIN2+ will be estimated directly using the women who test positive with a particular screening test. An unbiased estimate of NPV will be obtained by using only results for the 5% of women who are negative for the three screening tests who are randomly selected to receive colposcopy and a minimum of two biopsies. Methods that account for verification-biased sampling will be used to obtain unbiased estimates of sensitivity and specificity for CIN2+ detection.25 A method developed by Leisenring et.al. 26 will be used to test for significant differences in PPV and NPV.

ELIGIBILITY:
Inclusion Criteria:

* Women between 30 and 59 years of age

Exclusion Criteria:

* Pregnancy at the time of colposcopy/biopsy
* Hysterectomy with surgically absent cervix
* HPV test in the last 5 years independently of negative or positive result
* Previous cervical cancer diagnosis or treatment in the last 5 years
* Lack of willingness or capacity to provide informed consent

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender women
Enrollment: 10000 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 12 months, non-randomized
  Proportion of true CIN2+ positive cases based on biopsy, detected by AVE compared to VIA.
Positive Predictive Value (PPV) | 12 months, non-randomized
  Proportion of participants with AVE positive tests that have cervical precancer based on biopsy compared to those with positive VIA positive tests

CONTACTS AND LOCATIONS:
Overall Officials: Karla Alfaro, MD, Principal Investigator — Basic Health International; David Levitz, PhD, Principal Investigator — DL Analytics
Locations (1):
- Ministerio de Salud, San Salvador, El Salvador

REFERENCES:
- [Background] Rao DW, Bayer CJ, Liu G, Chikandiwa A, Sharma M, Hathaway CL, Tan N, Mugo N, Barnabas RV. Modelling cervical cancer elimination using single-visit screening and treatment strategies in the context of high HIV prevalence: estimates for KwaZulu-Natal, South Africa. J Int AIDS Soc. 2022 Oct;25(10):e26021. doi: 10.1002/jia2.26021. PMID 36225139
- [Background] Parham GP, Egemen D, Befano B, Mwanahamuntu MH, Rodriguez AC, Antani S, Chisele S, Munalula MK, Kaunga F, Musonda F, Malyangu E, Shibemba AL, de Sanjose S, Schiffman M, Sahasrabuddhe VV. Validation in Zambia of a cervical screening strategy including HPV genotyping and artificial intelligence (AI)-based automated visual evaluation. Infect Agent Cancer. 2023 Oct 16;18(1):61. doi: 10.1186/s13027-023-00536-5. PMID 37845724
- [Background] Hull R, Mbele M, Makhafola T, Hicks C, Wang SM, Reis RM, Mehrotra R, Mkhize-Kwitshana Z, Kibiki G, Bates DO, Dlamini Z. Cervical cancer in low and middle-income countries. Oncol Lett. 2020 Sep;20(3):2058-2074. doi: 10.3892/ol.2020.11754. Epub 2020 Jun 19. PMID 32782524
- [Background] Desai KT, Befano B, Xue Z, Kelly H, Campos NG, Egemen D, Gage JC, Rodriguez AC, Sahasrabuddhe V, Levitz D, Pearlman P, Jeronimo J, Antani S, Schiffman M, de Sanjose S. The development of "automated visual evaluation" for cervical cancer screening: The promise and challenges in adapting deep-learning for clinical testing: Interdisciplinary principles of automated visual evaluation in cervical screening. Int J Cancer. 2022 Mar 1;150(5):741-752. doi: 10.1002/ijc.33879. Epub 2021 Dec 6. PMID 34800038
- [Background] Xue Z, Novetsky AP, Einstein MH, Marcus JZ, Befano B, Guo P, Demarco M, Wentzensen N, Long LR, Schiffman M, Antani S. A demonstration of automated visual evaluation of cervical images taken with a smartphone camera. Int J Cancer. 2020 Nov 1;147(9):2416-2423. doi: 10.1002/ijc.33029. Epub 2020 May 19. PMID 32356305
- [Background] Ebrahimi N, Yousefi Z, Khosravi G, Malayeri FE, Golabi M, Askarzadeh M, Shams MH, Ghezelbash B, Eskandari N. Human papillomavirus vaccination in low- and middle-income countries: progression, barriers, and future prospective. Front Immunol. 2023 May 12;14:1150238. doi: 10.3389/fimmu.2023.1150238. eCollection 2023. PMID 37261366
- [Background] Desai KT, Ajenifuja KO, Banjo A, Adepiti CA, Novetsky A, Sebag C, Einstein MH, Oyinloye T, Litwin TR, Horning M, Olanrewaju FO, Oripelaye MM, Afolabi E, Odujoko OO, Castle PE, Antani S, Wilson B, Hu L, Mehanian C, Demarco M, Gage JC, Xue Z, Long LR, Cheung L, Egemen D, Wentzensen N, Schiffman M. Design and feasibility of a novel program of cervical screening in Nigeria: self-sampled HPV testing paired with visual triage. Infect Agent Cancer. 2020 Oct 14;15:60. doi: 10.1186/s13027-020-00324-5. eCollection 2020. PMID 33072178
- [Background] de Sanjose S, Perkins RB, Campos N, Inturrisi F, Egemen D, Befano B, Rodriguez AC, Jeronimo J, Cheung LC, Desai K, Han P, Novetsky AP, Ukwuani A, Marcus J, Ahmed SR, Wentzensen N, Kalpathy-Cramer J, Schiffman M; PAVE Study Group. Design of the HPV-automated visual evaluation (PAVE) study: Validating a novel cervical screening strategy. Elife. 2024 Jan 15;12:RP91469. doi: 10.7554/eLife.91469. PMID 38224340
- [Background] Hu L, Bell D, Antani S, Xue Z, Yu K, Horning MP, Gachuhi N, Wilson B, Jaiswal MS, Befano B, Long LR, Herrero R, Einstein MH, Burk RD, Demarco M, Gage JC, Rodriguez AC, Wentzensen N, Schiffman M. An Observational Study of Deep Learning and Automated Evaluation of Cervical Images for Cancer Screening. J Natl Cancer Inst. 2019 Sep 1;111(9):923-932. doi: 10.1093/jnci/djy225. PMID 30629194

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT06815939/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT06815939/ICF_001.pdf